CLINICAL TRIAL: NCT05584267
Title: Multi-omics Evaluation System and Preferred Mode of Immune Treatment of Brain Metastasis of Lung Cancer Combined With Large-segmentation Precision Radiotherapy
Brief Title: Immune Treatment of Brain Metastasis of Lung Cancer Combined With Large-segmentation Precision Radiotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Hunan Province Tumor Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RENO
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy; Drug Therapy; Immunotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cohort A (Active Comparator): Chemotherapy + immunotherapy; Every three weeks, up to four cycles of chemotherapy
  Interventions: Drug: Chemotherapy + immunotherapy
- cohort B (Experimental): Chemotherapy + immunotherapy; Once every three weeks, up to 4 cycles of chemotherapy; WBRT, 3 Gy/ time, 10 times in total
  Interventions: Radiation: radiotherapy; Drug: Chemotherapy + immunotherapy
- cohort C (Experimental): Chemotherapy + immunotherapy; Once every three weeks, up to 4 cycles of chemotherapy; HFRT, 10 Gy/ time, 3 times in total
  Interventions: Radiation: radiotherapy; Drug: Chemotherapy + immunotherapy

INTERVENTIONS:
Radiation: radiotherapy — Different cohorts received different doses of radiotherapy
  Arms: cohort B; cohort C
Drug: Chemotherapy + immunotherapy — Chemotherapy + immunotherapy

SUMMARY:
This is a prospective multicenter clinical study. This study aims to construct an auxiliary decision-making system for lung cancer immunotherapy combined with radiotherapy by fusing three modes of imagomics, clinicopathological features, and molecular pathological features.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age on day of signing informed consent
* Histopathology confirmed non-small cell lung cancer
* Asymptomatic brain metastases
* EGFR/ALK ROS1 driver gene mutation negative
* RECIST 1.1 based available assessment of lesions
* ECOG 0-1
* Brain metastases 1-4
* Single lesion ≤4cm

Exclusion Criteria:

* Patients with contraindication of chemotherapy Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-12-25 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Intracranial progression-free survival | up to 2 years from enrollment
  assessed according to the Response Evaluation Criteria in Solid Tumors RECIST Version 1.1, undergoing enhanced CT/MRI
sPFS | up to 2 years from enrollment
  assessed according to the Response Evaluation Criteria in Solid Tumors RECIST Version 1.1, undergoing enhanced CT/MRI

SECONDARY OUTCOMES:
Objective Response rate | up to 2 years from enrollment
  assessed according to the Response Evaluation Criteria in Solid Tumors RECIST Version 1.1, undergoing enhanced CT/MRI
overall survival | up to 2 years from enrollment
  the time from enrollment until death or the last follow-up
number of participants with treatment-related adverse events | up to 2 years from enrollment
  number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China